CLINICAL TRIAL: NCT02720263
Title: A Phase 1 Multiple Ascending Oral Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ASP4345 in Patients With Schizophrenia
Brief Title: A Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ASP4345 in Patients With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4345-CL-0002
Record Dates: First submitted 2016-03-22; First posted 2016-03-25 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; ASP4345
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Double-Blind ASP4345 Multiple Dose Levels (Experimental): ASP4345 will be administered orally as a single daily dose on days 1 through 14 with water. On days 1, 7, and 14, ASP4345 will be administered under fasting conditions. On days 2-6 and 8-13, ASP4345 will be administered under fed conditions.
  Interventions: Drug: ASP4345
- Double-Blind Placebo Multiple Dose (Placebo Comparator): Matching placebo capsules will be administered orally as a single daily dose on days 1 through 14 with water. On days 1, 7, and 14, matching placebo capsules will be administered with food. On days 2-6 and 8-13, matching placebo will be administered under fed conditions.
  Interventions: Drug: Matching Placebo
- Open-Label ASP4345 (Experimental): ASP4345 will be administered orally as a single daily dose on days 1 through 14 with water. On days 1, 7, and 14, ASP4345 will be administered with food. On days 2-6 and 8-13, ASP4345 will be administered under fed conditions. This is an optional cohort where subjects will be enrolled to further characterize pharmacodynamics in the event a higher sample size is necessary to determine changes in electrophysiological biomarkers.
  Interventions: Drug: ASP4345

INTERVENTIONS:
Drug: ASP4345 — Oral
  Arms: Double-Blind ASP4345 Multiple Dose Levels; Open-Label ASP4345
Drug: Matching Placebo — Oral
  Arms: Double-Blind Placebo Multiple Dose

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of multiple ascending oral doses of ASP4345 in patients with schizophrenia. In addition, this study will evaluate the pharmacokinetics of multiple ascending oral doses of ASP4345 in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a diagnosis of schizophrenia or schizoaffective disorder according to the Diagnostic and Statistical Manual of Mental Disorders, 5th edition criteria.
* A patient is considered operationally stable if the patient has a low to moderate positive symptoms score and moderate negative symptom score on the Positive and Negative Syndrome Scale (PANSS): No more than moderate rating on more than 2 PANSS items P1, P2, P3, P5, P6 (positive symptom section); No more than moderate severity rating for the negative items, N1, N2, N3, N4, N5, N6, N7 (negative symptom section); total PANSS score no more than 80.
* Patient must be in ongoing maintenance antipsychotic therapy other than clozapine (oral or depot), on a stable (≤ 25% change in dose) medication treatment regimen (approved oral or depot formulations of risperidone, quetiapine, olanzapine, ziprasidone, brexpiprazole, aripiprazole, paliperidone or lurasidone) for ≥ 2 months for oral formulations or ≥ 3 months for depot formulations prior to screening, including concomitant psychotropic medications, such as, trazodone and zolpidem for sleep.
* Patient has a body mass index (BMI) range of 18.5 to 40.0 kg/m2, inclusive, and weighs at least 50 kg at screening.
* Female patient must be of nonchildbearing potential:

  * Postmenopausal (defined as at least 1 year without any menses) prior to screening, or
  * Documented surgically sterile (at least 1 month prior to screening defined as hysterectomy, bilateral salpingectomy and/or bilateral oophorectomy)
* Female patient must not donate ova starting at screening and throughout the study period, and for 28 days after the final study drug administration.
* Male patient and their female spouse/partners who are of childbearing potential must be using 2 forms of highly effective birth control† (1 of which must be a barrier method‡) starting at screening and continue throughout the study period and for 90 days after the final study drug administration.

  †Highly effective forms of birth control include:
  * Consistent and correct usage of established oral contraception
  * Injected or implanted hormonal methods of contraception
  * Established intrauterine device or intrauterine system
  * Bilateral tubal ligation
  * Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments and complies with the preferred and usual lifestyle of the patient.

    ‡Barrier methods of birth control include:
  * Condom with spermicidal foam/gel/film/cream/suppository
  * Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository
* Male patient must not donate sperm starting at screening and throughout the study period and for 90 days after the final study drug administration.
* Patient agrees not to participate in another interventional study while participating in the present study, defined as signing the informed consent form until the end of study visit (ESV).
* Patient has a negative urine drug screen for drugs of abuse at screening and check in.

Exclusion Criteria:

* Female patient who has been pregnant within 6 months prior to screening assessment or breastfeeding within 3 months prior to screening.
* Patient has a known or suspected hypersensitivity to ASP4345 or any components of the formulation used.
* Patient has had previous exposure with ASP4345.
* Patient has a history of suicide attempt or suicidal behavior within 2 years prior to screening. Any suicidal ideation that meets criteria at a level of 4 or 5 by using C-SSRS within the last 3 months or who is at significant risk to commit suicide at screening or at admission to the clinical unit (day 2) will be excluded.
* Patient has any clinically significant liver chemistry test result aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), gamma glutamyl transferase, total bilirubin (TBL) or a result > than 1.5 times above the ULN at screening or at admission to the clinical unit (day 2). In such a case, the assessment may be repeated once.
* Patient has any history of allergic conditions deemed clinically significant.
* Patient has any history or evidence of any clinically significant cardiovascular, gastrointestinal endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric (other than schizophrenia or schizoaffective disorder), renal and/or other major disease or malignancy. Patient has any condition, which, makes the patient unsuitable for clinical study participation.
* Patient has been diagnosed with moderate or severe tardive dyskinesia, bipolar disorder, major depressive disorder, personality disorders, neuroleptic malignancy syndrome or anxiety disorder.
* Patient has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (noncutaneous) infection within 1 week prior to admission to the clinical unit (day 2).
* Patient has any clinically significant abnormality at screening or at admission to the clinical unit (day 2).
* Patient has a mean pulse < 40 or > 100 bpm; mean systolic blood pressure (SBP) > 160 mmHg; mean diastolic blood pressure (DBP) > 90 mmHg (vital signs measurements taken in triplicate after patient has been resting in supine position for 5 minutes; pulse will be measured automatically) at screening or at admission to the clinical unit (day 2). If the mean blood pressure exceeds the limits above, 1 additional triplicate can be taken on day 2.
* Patient has a mean QTcF > 440 msec (for male patients) and > 460 msec (for female patients) at screening or at admission to the clinical unit (day 2). If the mean QTcF exceeds the limits above, 1 additional triplicate ECG can be taken on day 2.
* Patient uses any prescribed or nonprescribed drugs (including vitamins, natural and herbal remedies, e.g., Valerian) in the 2 weeks prior to study drug administration, except for:

  1. Approved antipsychotics (risperidone, quetiapine, olanzapine, ziprasidone, brexpiprazole, aripiprazole, paliperidone or lurasidone), or
  2. Approved intermittent use of trazodone or zolpidem (no less than 12 hours prior to dosing), or
  3. Approved use of concomitant medication for the treatment of hypertension, hyperlipidemia or diabetes mellitus, or
  4. Occasional use of acetaminophen (up to 2 g/day).
* Patient has a history of consuming more than 14 units of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical/substance abuse within past 2 years prior to screening (Note: 1 unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits/hard liquor) or the patient tests positive for alcohol or drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and opiates) at screening or at admission to the clinical unit (day 2). A patient with a positive result for benzodiazepines may be included in this clinical study, if the result can be explained by the use of permitted concomitant medication.
* Patient has used any strong CYP3A inhibitors (e.g., but not limited to: boceprevir, clarithromycin, conivaptan, indinavir, itraconazole, ketoconazole, lopinavir/ritonavir, mibefradil, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telaprevir, telithromycin, voriconazole) and/or has consumed grapefruit, grapefruit containing products, Seville orange or Seville orange containing products within 72 hours prior to admission to the clinical unit (day 2).
* Patient has used any strong or moderate CYP2D6 inhibitors (e.g., but not limited to: bupropion, fluoxetine, paroxetine, quinidine, cinacalcet, duloxetine, terbinafine) within 72 hours prior to admission to the clinical unit (day 2).
* Patient regularly uses any inducer of metabolism (e.g., but not limited to: barbiturates, rifampin, St. John's Wort) in the 1 month prior to admission to the clinical unit (day 2).
* Patient has used any drugs of abuse within 3 months prior to admission to the clinical unit (day 2).
* Patient has had significant blood loss, donated 1 unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to admission to the clinical unit (day 2).
* Patient has a positive serology test for hepatitis B surface antigen (HBsAg), hepatitis A virus (HAV) antibodies (immunoglobulin M [IgM]), hepatitis C virus (HCV) antibodies, or human immunodeficiency virus (HIV) antibodies type 1 or 2 at screening.
* Patient has participated in any clinical study or has been treated with any investigational drugs within 28 days or 5 half lives whichever is longer, prior to screening.
* Patient is an employee of the Astellas Group or Contract Research Organization (CRO) involved in the clinical study.
* Patient who has had electroconvulsive therapy within the 6 months prior to screening.
* Patient has a history of seizures or of a condition with risk of seizures; as an exception, a history of 1 febrile seizure in childhood will not exclude a patient.
* Patient has a history of head injury with clinically significant sequelae.
* Patient experienced an acute exacerbation of schizophrenia requiring hospitalization within the last 3 months.
* Patient experienced an acute exacerbation of schizophrenia requiring increase in antipsychotic medication (with reference to drug or dose) within the last 4 weeks.
* Patient has hearing loss, is unable to detect 1000 Hz tones presented at 40 dB.
* Patient has a hairstyle that would interfere with electroencephalogram (EEG) recording quality.
* Patient has a history of spine surgery (with intact dura mater) in the past year and/or a history of brain and/or spinal cord injury.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-03-28 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed as nature, frequency and severity of adverse events | Up to Day 21
Change from baseline in supine blood pressure as a measure of safety and tolerability | Baseline and Day 21
Change from baseline in pulse as a measure of safety and tolerability | Baseline and Day 21
Change from baseline in oral body temperature as a measure of safety and tolerability | Baseline and Day 21
Safety and tolerability assessed by an orthostatic challenge test | Up to Day 14
  Incidence of positive orthostatic challenge tests will be summarized.
Number of participants with abnormal laboratory values and/or adverse events related to treatment | Up to Day 21
  Clinical laboratory tests include hematology, biochemistry and urinalysis.
Safety and tolerability assessed by routine 12-lead electrocardiogram (ECG) | Up to Day 18
  The overall interpretation of 12-lead electrocardiogram (ECG) results (normal, abnormal not clinically significant and abnormal clinically significant) will be summarized.
Safety and tolerability assessed by continuous 12-lead ECG recording | Up to Day 14
  ECGs will be collected using a 12-lead ECG continuous monitoring system which records continuous digital data.
Safety and tolerability assessed by abuse liability using an Addiction Research Center Inventory (ARCI-49) | Up to Day 17
  ARCI-49 is a 49-item short form standardized questionnaire for abuse potential liability.
Safety and tolerability assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to Day 18
  The C-SSRS is a scale that assesses the full spectrum of suicidality: suicidal ideation, intensity of ideation, suicidal behaviors and actual attempts.
Safety and tolerability assessed by Bond-Lader Visual Analog Scale (VAS) | Up to Day 17
  The VAS will be used to rate patients' feelings in terms of 16 dimensions. The dimensions will be presented as 100 mm lines, the 2 extremes of the emotion (i.e., alert - drowsy) written at each end.
Safety and tolerability assessed by metabolic syndrome: weight circumference | Up to Day 14
Safety and tolerability assessed by metabolic syndrome: cholesterol | Up to Day 21
Safety and tolerability assessed by metabolic syndrome: triglycerides | Up to Day 21
Safety and tolerability assessed by metabolic syndrome: glucose level | Up to Day 21
Safety and tolerability assessed by weight | Up to Day 14
Safety and tolerability assessed by movement disorder: Abnormal Involuntary Movement Scale (AIMS) | Up to Day 14
  The AIMS is a checklist and uses a 5-point rating scale for recording scores for 7 body areas: face, lips, jaw, tongue, upper extremities, lower extremities and trunk.
Safety and tolerability assessed by movement disorder: Simpson Angus Scale (SAS) | Up to Day 14
  The SAS is a 10-item scale used to rate adverse neurological effects of antipsychotic medications more broadly. Each item is rated from 0 to 4 and a total score will be obtained.
Safety and tolerability assessed by movement disorder: Barnes Akathisia Rating Scale (BARS) | Up to Day 14
  The BARS is a rating scale used to assess the severity of drug-induced akathisia.
Pharmacokinetics of ASP4345 and its metabolites, if necessary (plasma): tlag | Day 1
  Time prior to the time corresponding to the first measurable (nonzero) concentration (tlag)
Pharmacokinetics of ASP4345 and its metabolites, if necessary (plasma): tmax | Day 1 and Day 14
  Time of maximum concentration (tmax)
Pharmacokinetics of ASP4345 and its metabolites, if necessary (plasma): Cmax | Day 1 and Day 14
  Maximum concentration (Cmax)
Pharmacokinetics of ASP4345 and its metabolites, if necessary (plasma): AUCtau | Day 1 and Day 14
  Area under the concentration-time curve from the time of dosing to the start of the next dosing interval (AUCtau)
Pharmacokinetics of ASP4345 and its metabolites, if necessary (plasma): Ctrough | Days 2 through 14
  Concentration immediately prior to dosing at multiple dosing (Ctrough)
Pharmacokinetics of ASP4345 and its metabolites, if necessary (plasma): t1/2 | Day 14
  Terminal elimination half-life (t1/2)
Pharmacokinetics of ASP4345 and its metabolites, if necessary (plasma): MRTinf | Day 14
  Mean residence time extrapolated to time infinity (MRTinf)
Pharmacokinetics of ASP4345 and its metabolites, if necessary (plasma): terminal elimination rate constant | Day 14
Pharmacokinetics of ASP4345 and its metabolites, if necessary (plasma): Vz/F | Day 14
  Apparent volume of distribution during the terminal elimination phase after single extravascular dosing (Vz/F)
Pharmacokinetics of ASP4345 and its metabolites, if necessary (plasma): CL/F | Day 14
  Apparent total systemic clearance after extravascular dosing (CL/F)
Pharmacokinetics of ASP4345 and its metabolites, if necessary (plasma): Rac(AUC) | Day 14
  Accumulation index area under the concentration-time curve (Rac(AUC))
Pharmacokinetics of ASP4345 and its metabolites, if necessary (plasma): PTR | Day 14
  Peak trough ratio (PTR)
Pharmacokinetics of ASP4345 and its metabolites, if necessary (urine): Aetau | Day 14
  Cumulative amount of study drug excreted into urine from the time of dosing to the start of the next dosing interval (Aetau)
Pharmacokinetics of ASP4345 and its metabolites, if necessary (urine): Aetau% | Day 14
  Percentage of study drug dose excreted into urine from the time of dosing to the start of the next dosing interval (Aetau%)
Pharmacokinetics of ASP4345 and its metabolites, if necessary (urine): CLR | Day 14
  Renal clearance (CLR)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Clinical Pharmacology and Exploratory Development
Locations (1):
- Site US10001, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Desai A, Benner L, Wu R, Gertsik L, Maruff P, Light GA, Uz T, Marek GJ, Zhu T. Phase 1 randomized study on the safety, tolerability, and pharmacodynamic cognitive and electrophysiological effects of a dopamine D1 receptor positive allosteric modulator in patients with schizophrenia. Neuropsychopharmacology. 2021 May;46(6):1145-1151. doi: 10.1038/s41386-020-00908-0. Epub 2020 Nov 17. PMID 33203954
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/study.aspx?ID=403